CLINICAL TRIAL: NCT02308449
Title: Effects of Endogenous Iron Status and Intravenous Iron on Human Skeletal Muscle Metabolism at Rest and During Exercise
Brief Title: Iron Status and Human Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13/SC/0439
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iron-deficient, given placebo (Placebo Comparator): Iron-deficient participants given an infusion of sodium chloride at conclusion of baseline experimental visit
  Interventions: Drug: Sodium chloride (placebo)
- Iron-deficient, given iron (Active Comparator): Iron-deficient participants given an infusion of ferric carboxymaltose at conclusion of baseline experimental visit
  Interventions: Drug: Ferric carboxymaltose
- Iron-replete, given placebo (Placebo Comparator): Iron-replete participants given an infusion of sodium chloride at conclusion of baseline experimental visit
  Interventions: Drug: Sodium chloride (placebo)
- Iron-replete, given iron (Active Comparator): Iron-deficient participants given an infusion of ferric carboxymaltose at conclusion of baseline experimental visit
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Infusion of 15 mg/kg (up to maximum 1000 mg) ferric carboxymaltose in 250 mL 0.9% sodium chloride
  Other Names: Ferinject
  Arms: Iron-deficient, given iron; Iron-replete, given iron
Drug: Sodium chloride (placebo) — Infusion of 250 mL 0.9% sodium chloride
  Other Names: Normal saline
  Arms: Iron-deficient, given placebo; Iron-replete, given placebo

SUMMARY:
Iron deficiency is common in cardiorespiratory diseases and appears to contribute to a worse outcome. This human physiology study will examine the extent to which human skeletal muscle metabolism and exercise physiology are impaired by iron deficiency.

DETAILED DESCRIPTION:
This is a prospective double-blind randomised controlled study of the effect of endogenous iron status on skeletal muscle metabolism and exercise physiology. 32 healthy volunteers will take part, half of whom will be iron-deficient. The study involves a screening visit and two half-day visits during which assessments are performed. 50% of each group will be randomised to receive iron-repletion with ferric carboxymaltose at the end of the first experimental visit before returning to repeat identical assessments around one week later. This approach will make it possible to explore whether baseline differences in skeletal muscle metabolism are explained by differences in iron status per se, whilst controlling for any learning effect during participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Men and women aged 18 years or older and generally in good health
* For iron-deficient volunteers: ferritin ≤ 15 microg/L and transferrin saturation < 16%
* For iron-replete volunteers: ferritin ≥ 20 microg/L and transferrin saturation ≥ 20%

Exclusion Criteria:

* Haemoglobin < 8.0 g/dL
* Haemoglobinopathy
* Iron overload, defined as ferritin > 300 microg/L
* Hypoxaemia (SpO2 < 94%) or significant co-morbidity that may affect haematinics, metabolic or ventilatory responses
* Iron supplementation or blood transfusion within the previous 6 weeks
* Pregnancy or breast feeding
* Inability to exercise isolated calf muscle using a pedal or on a bicycle ergometer
* Contraindication to magnetic resonance spectroscopy exposure such as metallic implant
* Contraindication to receiving intravenous ferric carboxymaltose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Phosphocreatine depletion during small muscle mass exercise | 36 minute long graded exercise test; performed at baseline and follow-up visits (approximately a week apart)
  Degree of phosphocreatine depletion during graded exercise of calf muscle assessed using magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Cardiopulmonary exercise test performance | Hour long graded exercise test; performed at baseline and follow-up visits (approximately a week apart)
  Blood lactate and cardiorespiratory parameters during moderate large skeletal muscle mass exercise, assessed with cardiopulmonary exercise testing
Muscle biopsy findings | Immediately before and immediately after hour long cardiopulmonary exercise test, performed at baseline and follow-up visits (approximately a week apart)
  Skeletal muscle characteristics, assessed by minimally-invasive muscle biopsy (not a compulsory part of the protocol)
Participant reported symptoms | At study screening visit compared to four weeks following infusion of iron or placebo
  Measures of fatigue, restless-legs syndrome and well-being assessed by self-reported questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Robbins, DPhil, Study Director — University of Oxford; Matthew C Frise, MRCP, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford OCMR & CCRF, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Formenti F, Constantin-Teodosiu D, Emmanuel Y, Cheeseman J, Dorrington KL, Edwards LM, Humphreys SM, Lappin TR, McMullin MF, McNamara CJ, Mills W, Murphy JA, O'Connor DF, Percy MJ, Ratcliffe PJ, Smith TG, Treacy M, Frayn KN, Greenhaff PL, Karpe F, Clarke K, Robbins PA. Regulation of human metabolism by hypoxia-inducible factor. Proc Natl Acad Sci U S A. 2010 Jul 13;107(28):12722-7. doi: 10.1073/pnas.1002339107. Epub 2010 Jun 28. PMID 20616028
- [Background] Smith TG, Talbot NP, Privat C, Rivera-Ch M, Nickol AH, Ratcliffe PJ, Dorrington KL, Leon-Velarde F, Robbins PA. Effects of iron supplementation and depletion on hypoxic pulmonary hypertension: two randomized controlled trials. JAMA. 2009 Oct 7;302(13):1444-50. doi: 10.1001/jama.2009.1404. PMID 19809026
- [Background] Smith TG, Balanos GM, Croft QP, Talbot NP, Dorrington KL, Ratcliffe PJ, Robbins PA. The increase in pulmonary arterial pressure caused by hypoxia depends on iron status. J Physiol. 2008 Dec 15;586(24):5999-6005. doi: 10.1113/jphysiol.2008.160960. Epub 2008 Oct 27. PMID 18955380
- [Background] Smith TG, Brooks JT, Balanos GM, Lappin TR, Layton DM, Leedham DL, Liu C, Maxwell PH, McMullin MF, McNamara CJ, Percy MJ, Pugh CW, Ratcliffe PJ, Talbot NP, Treacy M, Robbins PA. Mutation of von Hippel-Lindau tumour suppressor and human cardiopulmonary physiology. PLoS Med. 2006 Jul;3(7):e290. doi: 10.1371/journal.pmed.0030290. PMID 16768548
- [Background] Finch CA, Gollnick PD, Hlastala MP, Miller LR, Dillmann E, Mackler B. Lactic acidosis as a result of iron deficiency. J Clin Invest. 1979 Jul;64(1):129-37. doi: 10.1172/JCI109431. PMID 447849
- [Result] Frise MC, Holdsworth DA, Johnson AW, Chung YJ, Curtis MK, Cox PJ, Clarke K, Tyler DJ, Roberts DJ, Ratcliffe PJ, Dorrington KL, Robbins PA. Abnormal whole-body energy metabolism in iron-deficient humans despite preserved skeletal muscle oxidative phosphorylation. Sci Rep. 2022 Jan 19;12(1):998. doi: 10.1038/s41598-021-03968-4. PMID 35046429